CLINICAL TRIAL: NCT06609655
Title: AgeTeQ Database Management Framework "Arts, Health and New Information and Communication Technologies"
Brief Title: AgeTeQ Database Management Framework
Status: Not yet recruiting | Type: Observational
Sponsor: Olivier Beauchet (Other Government)
Collaborators: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Responsible Party: Sponsor-Investigator, Olivier Beauchet, MD PhD, Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal
Organization: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Other Study IDs: 2025-227
Record Dates: First submitted 2024-09-18; First posted 2024-09-24 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Adults 18 Years and Older (no Other Exclusion Criteria)
Keywords: arts and health; telehealth
MeSH Terms: conditions — Arts syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- adults: Adults 18 years old and more, male and female, having participated in one research project and agreeing that data are integrated in the databank
  Interventions: Other: no intervention studied, it's a databank

INTERVENTIONS:
Other: no intervention studied, it's a databank — The AgeTeQ database "Arts, health and new information and communication technologies" has three objectives.
  The first is to preserve the data collected as part of the research projects carried out by the AgeTeQ laboratory.
  The second objective of the database is to use the information provided by the recorded data to fuel reflection, test new research hypotheses and thus open up new avenues of research for the Arts, Health and New Information and Communication Technologies research team.
  The third objective is to share the AgeTeQ database with the scientific community on a non-commercial basis, to improve access to data on the themes of arts, health and new technologies, and to increase knowledge and enable the development of research in these fields.

SUMMARY:
The AgeTeQ "Arts, health and new information and communication technologies (NICTs)" laboratory database contains all the clinical and paraclinical data of participants in clinical research projects carried out by the AgeTeQ laboratory on the themes of the arts, and/or health, and/or NICTs.

The database can thus contain quantitative data (i.e. non-invasive measurements taken with questionnaires or measuring devices providing numerical values such as blood pressure, heart rate or electrical activity of the brain, etc.) and qualitative data (i.e. extracted from a verbatim in the context of guided interviews) from participants in the above-mentioned clinical research projects. These data can take the form of spreadsheets containing numerical values, written documents such as verbatims, and audio or video recordings.

ELIGIBILITY:
Inclusion Criteria:

* Had participate to a previous research project managed by the administrator of the databank
* Agreed to integrated the databank

Exclusion Criteria:

* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The bank will be set up within the framework of various research projects of the databank administrator.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2044-10 (Estimated); Study Completion 2044-10 (Estimated)

PRIMARY OUTCOMES:
Preserve the data collected as part of the research projects carried out by the AgeTeQ laboratory | 20 years
  To centralized harmonize data from different protocols in the field of interest
Analyze the data collected as part of the research projects carried out by the AgeTeQ laboratory | 20 years
  To analyze data to fuel reflection, test new research hypotheses and thus open up new avenues of research for the Arts, Health and New Information and Communication Technologies
Share the data collected as part of the research projects carried out by the AgeTeQ laboratory | 20 years
  To improve access to data on the themes of arts, health and new technologies, and to increase knowledge and enable the development of research in these fields.

IPD SHARING:
Plan to Share IPD: Undecided